CLINICAL TRIAL: NCT00372775
Title: A Phase 2 Efficacy And Safety Study Of SU011248 In Patients With Non-Small Cell Lung Cancer And Brain Metastases
Brief Title: Study Tests The Safety And Effectiveness Of SU011248 In Patients With Non-Small Cell Lung Cancer Having Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181092
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: brain metastases; Sunitinib; Phase 2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental)
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 37.5 mg daily by oral capsule in a continuous regimen until progression or unacceptable toxicity
  Other Names: Sutent

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of SU011248 in patients with non-small cell lung cancer with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologically proven brain metastases secondary to non-small cell lung cancer
* Received previous whole brain radiation therapy and none, 1 or 2 prior systemic therapy for the treatment of advanced/metastatic non-small cell lung cancer

Exclusion Criteria:

* Patients with brainstem lesions, spinal cord compression. carcinomatous meningitis, or leptomeningeal disease.
* Brain metastases >4 cm in any linear direction
* Intracranial or intratumoral hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (13):
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Cocoa Beach, Florida
  - Pfizer Investigational Site, Merritt Island, Florida
  - Pfizer Investigational Site, Titusville, Florida
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Basking Ridge, New Jersey
  - Pfizer Investigational Site, Commack, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Sayre, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Round Rock, Texas
- France (4):
  - Pfizer Investigational Site, Pessac, Be1 04495
  - Pfizer Investigational Site, Saint-Priest-en-Jarez, France
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Toulouse
- Italy (4):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Orbassano (TO)
  - Pfizer Investigational Site, Roma
- Spain (2):
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181092&StudyName=Study%20Tests%20The%20Safety%20And%20Effectiveness%20Of%20SU011248%20In%20Patients%20With%20Non-Small%20Cell%20Lung%20Cancer%20Having%20Brain%20Metastases

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Sunitinib 37.5 mg oral capsule daily
Period: Overall Study
Arm/Group | Sunitinib
Started | 66
Received Treatment | 64
Completed | 3
Not Completed | 63
Not completed — Adverse Event | 8
Not completed — Death | 15
Not completed — Objective progression or relapse | 30
Not completed — Global deterioration of health status | 6
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1
Not completed — Not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Age, Customized [Number; unit: Participants]
  Between 18 and 44 years | 4
  Between 45 and 64 years | 40
  >= 65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. Since day of first dose of medication and day criteria for progression were met, were each counted as a full day, 1 day was added to each calculation. PFS calculated as (first event date minus date of first dose of study medication plus 1) divided by 7.02. Used 7.02 days because it equals(=) 365 days per year divided by 52 weeks per year. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]).
Time Frame: Baseline, Day 1 of Week 5, 9, 17, 25, 33, and 41 to tumor progression or death (up to 1 year)
Population: Intent-to-treat (ITT): all participants enrolled in the study who received at least 1 dose of study medication.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Weeks | 9.4 [7.5 to 13.1]

2. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time from start of study treatment to first documentation of objective tumor progression. Tumor progression defined as greater than or equal to 20 percent (≥20%) increase in sum of longest dimensions of target lesions using as reference smallest sum of longest dimensions recorded since treatment started, or unequivocal progression of existing non-target lesions, or appearance of ≥1 new lesion, according to Response Evaluation Criteria in Solid Tumors (RECIST). TTP = (first event date minus date of first dose of study medication plus 1) divided by 7.02.
Time Frame: Baseline, Day 1 of Week 5, 9, 17, 25, 33, and 41 to tumor progression (up to 1 year)
Population: ITT
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Weeks | 15.1 [8.4 to 15.8]

3. Secondary Outcome: Time to Neurological Progression (TNP)
Description: Time in weeks between first date criteria for focal neurological deficit were met and date of first dose of medication. Criteria for focal neurological deficit included speech or language difficulties, vision changes, loss of coordination or fine motor control, and seizures. Since day of first dose of medication and day criteria for focal neurological deficit were met were each counted as a full day, 1 day was added to each calculation. TNP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7.02.
Time Frame: Baseline, Day 28 to focal neurological deficit (up to 1 year)
Population: ITT
Measure: Median (Full Range); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Weeks | 8.1 [0.4 to 58.8]

4. Secondary Outcome: Number of Participants With Objective Disease Response
Description: Objective disease response defined as participants with confirmed complete response (CR) or partial response (PR), according to Response Evaluation Criteria in Solid Tumors (RECIST). CR defined as disappearance of all target lesions. PR defined as ≥30% decrease in sum of longest dimensions of target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline and Day 1 of Week 5, 9, 17, 25, 33, 41, and 49
Population: ITT with measurable disease at baseline.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
Participants | 1
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 1.6, 95% CI 2-sided [0.0 to 8.8] — Two-Sided Confidence Interval (CI) from Exact Method using the F Distribution

5. Secondary Outcome: Time to Objective Intracranial Progression
Description: Time in weeks from start of study treatment to first documentation of objective intracranial tumor progression. Intracranial tumor progression defined as ≥25% increase from smallest size in sum of products of all enhancing tumors or appearance of any new tumor, according to World Health Organization (WHO) criteria. Since day of first dose of medication and day criteria for progression were met, were each counted as a full day, 1 day added to each calculation. Time to Objective Intracranial Progression = (first event date minus the date of first dose of study medication plus 1) divided by 7.02.
Time Frame: Baseline, Day 1 of Week 5, 9, 17, 25, 33, and 41 to intracranial tumor progression (up to 1 year)
Population: ITT
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Weeks | 15.4 [12.1 to 24.8]

6. Secondary Outcome: Number of Participants With Intracranial Objective Disease Response
Description: Intracranial objective disease response defined as participants with confirmed CR or PR, according to WHO criteria. CR defined as disappearance of all enhancing tumor. PR defined as a ≥50% reduction from baseline in sum of the products of all enhancing tumors.
Time Frame: Baseline and Day 1 of Week 5, 9, 17, 25, 33, 41, and 49
Population: ITT with measurable intracranial disease at baseline.
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 23
Participants | 1
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; ORR (percent) = 4.3, 95% CI 2-sided [0.1 to 21.9] — Two-Sided CI from Exact Method using the F Distribution

7. Secondary Outcome: Duration of Response (DR)
Description: DR defined as difference in weeks between first date criteria for progression occurred, or participant died due to any cause and first date that criteria for a PR or CR were met and subsequently confirmed ≥4 weeks later. Since day criteria for PR or CR were met and first day criteria for progression occurred (or participant died) were each counted as a full day, 1 day was added to each calculation. DR (in weeks) calculated as (first date of PD or death minus first date of CR or PR that was subsequently confirmed plus 1) divided by 7.02.
Time Frame: Day 7 of Week 4 and every 4 weeks up to 1 year
Population: ITT. DR only calculated for the subgroup of participants with an objective tumor response.
Measure: Number; unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 1
Weeks
  Overall | 32.1
  Intracranial | 8.26

8. Secondary Outcome: Overall Survival (OS)
Description: OS calculated as: (date of death minus date of first dose plus 1)divided by 30.4.
Time Frame: Baseline until death (up to 1 year)
Population: ITT. In the absence of confirmation of death, survival time was censored to last date of known contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Months | 5.8 [3.1 to 8.2]

9. Secondary Outcome: Percentage of Participants Surviving at 1 Year
Description: Percentage of those surviving at end of 1 year from the first dose of study treatment.
Time Frame: Year 1
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Percentage of participants | 23.4 [14.0 to 34.3]
Statistical Analysis 1: Comparison: Sunitinib; Test type: Superiority or Other; Percentage = 23.4, 95% CI 2-sided [14.0 to 34.3] — Probability of survival along with the corresponding 2-sided confidence interval for the log [-log(one-year survival rate)] calculated using a normal approximation and then back transformed to give a confidence interval for the one-year survival

10. Secondary Outcome: Number of Deaths Due to Intracranial Versus Systemic Progression
Description: Number of deaths determined to be intracranial versus systemic progression, according to investigators'assessment.
Time Frame: Baseline until death (up to 1 year)
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
Participants
  Systemic Progression | 48
  Intracranial Progression | 0

11. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy/National Comprehensive Cancer Network (FACT/NCCN) Lung Symptom Index (FLSI) Score
Description: Change from baseline in FLSI Score was calculated Day 1 of Cycle 2 to 13. Each cycle = 28 days. Scores ranged from 0 to 24. Higher scores indicated better outcomes.
Time Frame: Baseline, Day 1 of Week 5 and every 4 weeks to end of treatment (up to 1 year)
Population: ITT population of participants with post baseline patient-reported outcome data
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 45
Scores on a scale
  Baseline | 17.62 [16.01 to 19.22]
  Cycle 2, Day 1 | 0.52 [-0.89 to 1.92]
  Cycle 3, Day 1 | 1.11 [-0.57 to 2.80]
  Cycle 4, Day 1 | -0.48 [-2.94 to 1.99]
  Cycle 5, Day 1 | 0.64 [-1.03 to 2.31]
  Cycle 6, Day 1 | -0.63 [-2.30 to 1.05]
  Cycle 7, Day 1 | -0.66 [-2.14 to 0.82]
  Cycle 8, Day 1 | -0.66 [-1.76 to 0.45]
  Cycle 9, Day 1 | -0.60 [-2.55 to 1.35]
  Cycle10, Day 1 | -0.12 [-2.47 to 2.23]
  Cycle 11, Day 1 | -0.20 [-2.96 to 2.56]
  Cycle 12, Day 1 | -0.40 [-2.99 to 2.19]
  Cycle 13, Day 1 | -0.80 [-10.96 to 9.36]

12. Secondary Outcome: Change From Baseline in FACT/NCCN Brain Symptom Index (FBrSI) Score
Description: Change from baseline in FBrSI Score was calculated Day 1 of Cycle 2 to 13. Each cycle = 28 days. Scores ranged from 0 to 60. Higher scores indicated better outcomes.
Time Frame: Baseline, Day 1 of Week 5 and every 4 weeks to end of treatment (up to 1 year)
Population: ITT population of participants with post baseline patient-reported outcome data
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sunitinib
Number analyzed (Participants) | 45
Scores on a scale
  Baseline | 45.72 [43.52 to 47.92]
  Cycle 2, Day 1 | -1.25 [-2.84 to 0.34]
  Cycle 3, Day 1 | -0.58 [-3.52 to 2.37]
  Cycle 4, Day 1 | 0.66 [-2.34 to 3.65]
  Cycle 5, Day 1 | -1.87 [-5.21 to 1.46]
  Cycle 6, Day 1 | -1.92 [-5.96 to 2.12]
  Cycle 7, Day 1 | -2.00 [-5.80 to 1.80]
  Cycle 8, Day 1 | -0.73 [-4.46 to 2.99]
  Cycle 9, Day 1 | 0.40 [-3.07 to 3.88]
  Cycle 10, Day 1 | -1.83 [-5.11 to 1.45]
  Cycle 11, Day 1 | -1.50 [-6.09 to 3.09]
  Cycle 12, Day 1 | -4.50 [-15.33 to 6.33]
  Cycle 13, Day 1 | 1.21 [-8.77 to 11.20]

13. Secondary Outcome: Trough Plasma Concentrations (Ctrough) of Sunitinib
Description: A single blood sample (4 milliliters [mL]) collected pre-dose on Day 1 of Cycles 2, 3, and 4 to determine Ctrough of Sunitinib and its metabolite SU12662. Each cycle = 28 days. Ctrough defined as plasma concentration prior to study drug administration. Trough plasma concentrations were dose-corrected.
Time Frame: Day 1 of Week 5, 9, and 13
Population: ITT participants who had pharmacokinetic results for at least 1 day. Ctrough only calculated for subgroup of participants with observations (non-missing concentrations). n = number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
nanograms per milliliter (ng/mL)
  Cycle 2, Day 1 (n = 26) | 50.89 (20.47)
  Cycle 3, Day 1 (n = 21) | 46.27 (17.97)
  Cycle 4, Day 1 (n = 20) | 51.10 (23.13)

14. Secondary Outcome: Ctrough of Sunitinib Metabolite (SU012662)
Description: A single blood sample (4 mL) collected pre-dose on Day 1 of Cycles 2, 3, and 4 to determine Ctrough of Sunitinib and its metabolite SU12662. Each cycle = 28 days. Ctrough defined as plasma concentration prior to study drug administration. Trough plasma concentrations were dose-corrected.
Time Frame: Day 1 of Week 5, 9, and 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 64
ng/mL
  Cycle 2, Day 1 (n = 26) | 33.85 (17.64)
  Cycle 3, Day 1 (n = 21) | 28.45 (15.73)
  Cycle 4, Day 1 ( n = 20) | 28.91 (18.82)

15. Secondary Outcome: Correlation of Polymorphisms in c-Kit, Flt-3 and c-Fms With Blood Counts
Description: A blood sample (6mL) collected before treatment with Sunitinib and used to isolate deoxyribonucleic acid (DNA). These samples were not anonymized.
Time Frame: Day 1 prior to dosing
Population: ITT. c-Kit, Flt-3 and c-Fms with blood count samples collected; however, no statistical analyses performed since power was insufficient.
Measure: Number; unit: picograms per milliliter (pg/mL)
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Participants by Ribonucleic Acid (RNA) Expression Profile
Description: Tumor samples were not anonymized. RNA expression profile was to include colony-stimulating factor 1 receptor (CSF-1R), platelet-derived growth factor receptor alpha and beta (PDGFRalpha and PDGFRbeta), vascular endothelial growth factor (VEGF), VEGF-C, VEGF receptor 1, 2, and 3 (VEGFR1, VEGFR2, and VEGFR3), fibroblast growth factor (FGF), FMS-like tyrosine kinase 3 (FLT3), KIT (stem cell factor receptor), and RET (rearranged during transfection).
Time Frame: Day 1 of Week 1 and every 4 weeks up to 1 year
Population: ITT. Only 4 RNA samples were collected and no statistical analyses performed.
Measure: Number; unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

17. Secondary Outcome: PFS in Subgroups Defined by RNA Expression Profiles of Tumors
Description: PFS defined as time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was to be determined in subgroups defined by RNA Gene expression (CSF-1R, PDGFRalpha, PDGFRbeta, VEGF, VEGF-C, VEGFR1, VEGFR2, VEGFR3, FGF, FLT3, KIT, and RET) level (low/high relative to expression of Glyceraldehyde-3-Phosphate Dehydrogenase [GAPDH] reference gene). PFS calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7.02.
Time Frame: Day 1 of Week 1 and every 4 weeks up to 1 year
Population: ITT. Only 4 RNA samples were collected and no statistical analyses performed.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 34/64
Other Adverse Events (participants affected / at risk) | 63/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=64)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Disease progression (General disorders) | 13
General physical health deterioration (General disorders) | 2
Pyrexia (General disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Pulmonary function test decreased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Cerebellar syndrome (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=64)
Anaemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 14
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 11
Chest pain (General disorders) | 5
Fatigue (General disorders) | 23
Mucosal inflammation (General disorders) | 11
Pain (General disorders) | 5
Platelet count decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 16
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Dry skin (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.